CLINICAL TRIAL: NCT04897165
Title: Resilience Training With Mobile Heart Rate Variability Biofeedback for Work-related Stress in White-collar Employees and the Influence of the Lecture Format (Digital vs. Live) on Training Success
Brief Title: Resilience Training for Work-related Stress in Employees and the Influence of the Lecture Format on Training Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STM_05
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Work-Related Stress; Burnout
MeSH Terms: conditions — Occupational Stress; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resilience training with mobile HRV-BfB based on an e-learning approach (with digital lectures) (Experimental)
  Interventions: Other: Resilience training with mobile HRV-BfB based on an e-learning approach (with digital lectures)
- Resilience training with mobile HRV-BfB based on a blended learning approach (with live lectures) (Experimental)
  Interventions: Other: Resilience training with mobile HRV-BfB based on a blended learning approach (with live lectures)
- Waitlist controls (No Intervention)

INTERVENTIONS:
Other: Resilience training with mobile HRV-BfB based on an e-learning approach (with digital lectures) — A 4-week resilience training with a mobile HRV-BfB device. Participants received access to three online lectures at the start of the first, third, and forth training week (each lasting 60 minutes) to receive a theoretical base on resilience and to learn how to exercise with the HRV-BfB device. Participants were asked to exercise three times a day for 5 minutes in their occupational and leisure time with the HRV-BfB device.
  Arms: Resilience training with mobile HRV-BfB based on an e-learning approach (with digital lectures)
Other: Resilience training with mobile HRV-BfB based on a blended learning approach (with live lectures) — A 4-week resilience training with a mobile HRV-BfB device. Participants attended three live lectures at the start of the first, third, and forth training week (each lasting 90 minutes) to receive a theoretical base on resilience and to learn how to exercise with the HRV-BfB device. Participants were asked to exercise three times a day for 5 minutes in their occupational and leisure time with the HRV-BfB device.
  Arms: Resilience training with mobile HRV-BfB based on a blended learning approach (with live lectures)

SUMMARY:
A study to analyze the psychophysiological effects of a preventative, 4-week resilience training with mobile heart rate variability biofeedback (HRV-BfB) in a workplace setting and the influence of the lecture format (digital vs. live) on the training success.

DETAILED DESCRIPTION:
This was a three-arm, non-randomized, controlled trial to examine the effects of a preventative, 4-week resilience training with mobile HRV-BfB on work-related stress in white-collar employees. Participants were asked to exercise autonomously three times per day for five minutes with the mobile HRV-BfB device. They additionally attended three lectures at the beginning of the first, third, and forth week. The aim of the lectures was to mediate a theoretical knowledge and to prepare the participants for the autonomous training. To examine the potential influence of the lecture format, one group attended live lectures (blended learning condition) and one group received access to online lectures (e-learning condition). Results of study's outcome measures were compared with a waitlist control group. Outcome measures were assessed at baseline (T0), after the 4-week intervention (T1), and at 4-week follow-up (T2).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Employees of the company at which the study is conducted

Exclusion Criteria:

* Implanted pacemaker
* Medically diagnosed heart failure or arrhythmia
* Medically prescribed cardiac drugs (e.g., beta-blockers, diuretics, ACE inhibitors, calcium channel blockers, or antiarrhythmic agents)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
COPSOQ personal burnout after the intervention | After the 4-week intervention (T1)
  Personal burnout was assessed with the adapted German long version of the Copenhagen Psychosocial Questionnaire (COPSOQ) at T1. Six questions were answered on an ordinal scale, transformed to values ranging between 0=minimum value and 100=maximum value (higher values indicate a more severe burnout symptomatology) and averaged to obtain a scale score (0-100).

SECONDARY OUTCOMES:
Change in the COPSOQ scale personal burnout between baseline (T0) and 4-week follow-up (T2) | Baseline (T0) and 4-week follow-up (T2)
  Personal burnout was assessed with the adapted German long version of the Copenhagen Psychosocial Questionnaire (COPSOQ) at T0 and T2. Six questions were answered on an ordinal scale, transformed to values ranging between 0=minimum value and 100=maximum value (higher values indicate a more severe burnout symptomatology) and averaged to obtain a scale score (0-100).
Change in the COPSOQ scale subjective general health between baseline (T0), after the 4-week intervention (T1), and 4-week follow-up (T2) | Baseline (T0), after the 4-week intervention (T1), and 4-week follow-up (T2)
  The subjective general health was assessed with the adapted German long version of the Copenhagen Psychosocial Questionnaire (COPSOQ, originally derived from the EQ-5D) at T0, T1, and T2 (single question). The question was transformed to a scale ranging from 0=minimum value to 100=maximum value (lower values indicate a worse general health).
Change in the COPSOQ scale work-privacy conflict between baseline (T0), after the 4-week intervention (T1), and 4-week follow-up (T2) | Baseline (T0), after the 4-week intervention (T1), and 4-week follow-up (T2)
  Work-privacy conflict was assessed with the adapted German long version of the Copenhagen Psychosocial Questionnaire (COPSOQ) at T0 and T2. Five questions were answered on an ordinal scale, transformed to values ranging between 0=minimum value and 100=maximum value (higher values indicate a worse conflict) and averaged to obtain a scale score (0-100).
Change in the COPSOQ scale behavioral stress symptoms between baseline (T0), after the 4-week intervention (T1), and 4-week follow-up (T2) | Baseline (T0), after the 4-week intervention (T1), and 4-week follow-up (T2)
  Behavioral stress symptoms were assessed with the adapted German long version of the Copenhagen Psychosocial Questionnaire (COPSOQ) at T0 and T2. Eight questions were answered on an ordinal scale, transformed to values ranging between 0=minimum value and 100=maximum value (higher values indicate more severe stress symptoms) and averaged to obtain a scale score (0-100).
Change in the COPSOQ scale cognitive stress symptoms between baseline (T0), after the 4-week intervention (T1), and 4-week follow-up (T2) | Baseline (T0), after the 4-week intervention (T1), and 4-week follow-up (T2)
  Cognitive stress symptoms were assessed with the adapted German long version of the Copenhagen Psychosocial Questionnaire (COPSOQ) at T0 and T2. Four questions were answered on an ordinal scale, transformed to values ranging between 0=minimum value and 100=maximum value (higher values indicate more severe stress symptoms) and averaged to obtain a scale score (0-100).
Change in self-reported sleep quality between baseline (T0), after the 4-week intervention (T1), and 4-week follow-up (T2) | Baseline (T0), after the 4-week intervention (T1), and 4-week follow-up (T2)
  Self-reported sleep quality, latency, and sleep duration were assessed with the Pittsburgh Sleep Quality Index (PSQI) at T0, T1, and T2. Items were averaged to obtain values between 0 and 3 (higher values indicate a poorer sleep).
HRV analysis: Change in SDNN between baseline (T0) and after the 4-week intervention (T1) | Baseline (T0) and after the 4-week intervention (T1)
  Standard deviation of normal to normal (NN) intervals (ms). Recorded with the software InnerBalanceTM Trainer (HeartMath Deutschland GmbH, Germany) and analyzed with the software HRV-Scanner (BioSign GmbH, Germany).
HRV analysis: Change in RMSSD between baseline (T0) and after the 4-week intervention (T1) | Root mean square of successive differences (ms). Recorded with the software InnerBalanceTM Trainer (HeartMath Deutschland GmbH, Germany) and analyzed with the software HRV-Scanner (BioSign GmbH, Germany).
  Baseline (T0) and after the 4-week intervention (T1)
HRV analysis: Change in pNN50 between baseline (T0) and after the 4-week intervention (T1) | Baseline (T0) and after the 4-week intervention (T1)
  Percentage of successive NN intervals that differ from each other by more than 50 ms (%). Recorded with the software InnerBalanceTM Trainer (HeartMath Deutschland GmbH, Germany) and analyzed with the software HRV-Scanner (BioSign GmbH, Germany).
HRV analysis: Change in Baevsky's stress index between baseline (T0) and after the 4-week intervention (T1) | Baseline (T0) and after the 4-week intervention (T1)
  Baevsky's stress index is computed from the main characteristics of the inter-beat intervals histogram (mode value, mode amplitude, and variation range). Recorded with the software InnerBalanceTM Trainer (HeartMath Deutschland GmbH, Germany) and analyzed with the software HRV-Scanner (BioSign GmbH, Germany).
HRV analysis: Change in the degree of rhythmization between baseline (T0) and after the 4-week intervention (T1) | Baseline (T0) and after the 4-week intervention (T1)
  A measure that quantifies the respiratory sinus arrhythmia. Recorded with the software InnerBalanceTM Trainer (HeartMath Deutschland GmbH, Germany) and analyzed with the software HRV-Scanner (BioSign GmbH, Germany).
Training evaluation | After the 4-week intervention (T1)
  Participants rated the training success, integrability and the responding to questions and needs on a 5-point scale (1=positive, 5=negative).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Study Director — ARCIM Institute Academic Research in Complementary and Integrative Medicine
Locations (1):
- Arcim Institute, Filderstadt, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available, in addition to study protocol and informed consent form.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available upon publication for a duration of three months.
Access Criteria: The data will be made available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.

REFERENCES:
- [Derived] Vagedes J, Szoke H, Islam MOA, Sobh M, Kuderer S, Khazan I, Vagedes K. Mobile Heart Rate Variability Biofeedback for Work-Related Stress in Employees and the Influence of Instruction Format (Digital or Live) on Training Outcome: A Non-Randomized Controlled Trial. Appl Psychophysiol Biofeedback. 2025 Mar;50(1):79-93. doi: 10.1007/s10484-024-09671-0. Epub 2024 Nov 1. PMID 39485585